CLINICAL TRIAL: NCT04618874
Title: A RANDOMIZED TRIAL COMPARING PERCUTANEOUS ULTRASOUND-GUIDED NEEDLE ASPIRATION/BIOPSY WITH AND WITHOUT RAPID ON SITE EVALUATION IN PATIENTS WITH SUSPECTED SUPERFICIAL METASTASIS FROM LUNG CANCER
Brief Title: US NAB With ROSE Versus US FNAB With no ROSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 3866
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-02

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Rapid on-site cytological examination; Ultrasound-guided needle aspiration biopsy; Lung adenocarcinoma; Molecular profiling
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ROSE group (Experimental): Ultrasound-assisted percutaneous needle aspiration with rapid on-site evaluation
  Interventions: Diagnostic Test: Rapid on-site evaluation
- US NAB group (No Intervention): Ultrasound-assisted percutaneous needle aspiration without rapid on-site evaluation

INTERVENTIONS:
Diagnostic Test: Rapid on-site evaluation — Rapid on site evaluation performed with an MGG quick stain (Bio-Optica, Milano, Italy).
  Arms: ROSE group

SUMMARY:
This is an investigator-initiated, single center, controlled, randomized clinical trial with two parallel arms in a 1:1 ratio. The objective of the study is to systematically assess the influence of rapid on-site evaluation (ROSE) on the diagnostic yield for diagnosis and molecular profiling, as well as on the safety, of pulmonologist-performed ultrasound-assisted needle aspiration biopsy (US-NAB) of superficial lesions across different metastatic sites in a series of consecutive patients with suspect locally advanced or advanced lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Known/suspected lung cancer
* Presence of a suspected "superficial" metastasis at imaging studies (CT and/or PET)
* Indication to tissue sampling for diagnosis, staging and/or molecular profiling
* 18 years or older
* Provision of a written informed consent

Exclusion Criteria:

* Inability or unwillingness to consent
* Known bleeding disorder that cannot be sufficiently corrected with co-fact or fresh frozen plasma (FFP)
* Use of antiplatelet (excluded aspirin) or anticoagulant drugs that cannot be discontinued

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield for a tissue diagnosis | 20 days

SECONDARY OUTCOMES:
Diagnostic yield for cancer genotyping | 30 days
Diagnostic yield for PDL1 testing | 30 days
Complication rate | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Rocco Trisolini, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meena N, Bartter T. Ultrasound-guided Percutaneous Needle Aspiration by Pulmonologists: A Study of Factors With Impact on Procedural Yield and Complications. J Bronchology Interv Pulmonol. 2015 Jul;22(3):204-8. doi: 10.1097/LBR.0000000000000175. PMID 26165890
- [Background] Laursen CB, Naur TM, Bodtger U, Colella S, Naqibullah M, Minddal V, Konge L, Davidsen JR, Hansen NC, Graumann O, Clementsen PF. Ultrasound-guided Lung Biopsy in the Hands of Respiratory Physicians: Diagnostic Yield and Complications in 215 Consecutive Patients in 3 Centers. J Bronchology Interv Pulmonol. 2016 Jul;23(3):220-8. doi: 10.1097/LBR.0000000000000297. PMID 27454475
- [Background] Stigt JA, Oostdijk AH, Boers JE, van den Berg JW, Groen HJ. Percutaneous ultrasound-guided biopsies in the evaluation of thoracic tumours after PET-CT: a prospective diagnostic study. Respiration. 2012;83(1):45-52. doi: 10.1159/000330018. Epub 2011 Sep 16. PMID 21934274